CLINICAL TRIAL: NCT00421499
Title: Randomized Controlled, Parallel Group, Single Blinded, Phase 1 Study That Investigates the Effects of Regular Daily Intake of Small Amounts of Dark or White Chocolate on Blood Pressure in Elderly Individuals With Mild Hypertension
Brief Title: Effects of Cocoa Intake on Blood Pressure in Elderly Individuals With Mild Hypertension
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Cologne (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ECA-02-005
Record Dates: First submitted 2007-01-11; First posted 2007-01-12 (Estimated); Last update posted 2007-01-12 (Estimated); Status verified 2007-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension

INTERVENTIONS:
Drug: dark chocolate

SUMMARY:
Regular intake of cocoa-containing foods is linked to a considerably lower cardiovascular and all-cause mortality in observational studies. Short-term intervention studies indicate that high doses of cocoa improve endothelial function and reduce blood pressure (BP), but the clinical impact of long-term intake of small dietary amounts of cocoa on BP and the underlying BP lowering mechanisms are unclear. We hypothesized that cocoa consumption lowers blood pressure by augmentation of the circulating vasodilative nitric oxide (NO) pool due to the action of the cocoa polyphenols at the vascular endothelium.

To test this hypothesis, we will conduct a randomized single-blind, parallel group study in subjects with mild essential hypertension to evaluate the effects of polyphenol-rich dark chocolate versus polyphenol-free white chocolate on blood pressure and plasma levels of cocoa phenols, circulating bioactive nitric oxide, and plasma markers of oxidative stress. After a 7 day cocoa-free run-in period, 44 subjects will be 1:1 randomized to receive over 18 weeks daily doses of either dark chocolate (6.3 g per day with a total of 30 mg of polyphenols and 30 kcal) or polyphenol free white chocolate (5.6 g per day with 30 kcal, containing similar amounts of macronutrients, electrolytes and vitamins). Subjects will be counseled to maintain an isocaloric diet and to abstain from other cocoa products during the study. Blood pressure and plasma parameters will be assessed in each subject after the run-in period and after 6, 12, and 18 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 55 - 75 years in good general health with high normal blood pressure (between 130/80 and 140/90 mmHg) or mild hypertension (blood pressure between 140/90 and 160/100 mmHg)on no medication or nutritional supplements
* Non-manual workers with a household income > 20,000 €/year
* Normal plasma lipids (total plasma cholesterol < 6.18 mmol/L
* LDL < 4.11 mmol/L
* HDL > 0.9 mmol/L
* Triacylglycerols < 1.8 mmol/L) and normal plasma glucose (fasting plasma glucose 4.2-6.4 mmol/L).
* If a subject's blood pressure exceeds 170/100 mmHg on a single visit, the subject will be withdrawn from the study and referred to appropriate antihypertensive therapy.

Exclusion Criteria:

Subjects are excluded if they have:

* Cardiovascular diseases (other than hypertension)
* Diabetes mellitus
* Hyper-/dyslipidemia
* Gastrointestinal diseases
* Hepatic and renal disorders
* Pulmonary diseases
* Coagulopathy
* Cancer
* Psychiatric disorders
* Alcohol or drug dependence
* Seizure disorders
* History of organ transplantation
* Surgery within the last 12 months
* Positive tests for HIV, hepatitis B or C.

Subjects are excluded if they have:

* A body-mass index of more than 27.5 or less than 18.5 kg/m2
* Actively smoked tobacco within the last five years
* Regularly use medications
* Used any medication within the last two weeks before entry
* Use vitamin, mineral or polyphenol supplements or functional food.

Subjects will be excluded if they are unable to give informed consent for all procedures; or subjects who are not capable or willing to appear for controlling visits.

Ages: 55 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44
Dates: Start 2005-01; Study Completion 2005-05

PRIMARY OUTCOMES:
changes in systolic and diastolic blood pressure

SECONDARY OUTCOMES:
plasma levels of bioactive nitric oxide, 8-isoprostane, cocoa polyphenols

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Taubert, Principal Investigator — Department of Pharmacology, University of Cologne
Locations (1):
- Department of Pharmacology, University of Cologne, Cologne, Germany

REFERENCES:
- [Background] Taubert D, Berkels R, Roesen R, Klaus W. Chocolate and blood pressure in elderly individuals with isolated systolic hypertension. JAMA. 2003 Aug 27;290(8):1029-30. doi: 10.1001/jama.290.8.1029. No abstract available. PMID 12941673
- [Derived] Taubert D, Roesen R, Lehmann C, Jung N, Schomig E. Effects of low habitual cocoa intake on blood pressure and bioactive nitric oxide: a randomized controlled trial. JAMA. 2007 Jul 4;298(1):49-60. doi: 10.1001/jama.298.1.49. PMID 17609490